CLINICAL TRIAL: NCT00006445
Title: First and 2nd Trimester Evaluation of the Risk of Aneuploidy
Brief Title: Down Syndrome - Comparison of Screening Methods in the 1st and 2nd Trimesters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NICHD-0511; 1 RO1 HD37523
Record Dates: First submitted 2000-11-04; First posted 2000-11-06 (Estimated); Last update posted 2007-02-22 (Estimated); Status verified 2003-03

CONDITIONS: Down Syndrome; Chromosome Abnormalities
Keywords: Pregnancy; Ultrasound; Serum screen; Pregnancy associated plasma protein-A (PAPP-A); Free-beta human chorionic gonadotropin (FbhCG); Alpha fetoprotein; Unconjugated estriol; Inhibin-A; Down syndrome; Aneuploidy
MeSH Terms: conditions — Down Syndrome; Chromosome Aberrations; Aneuploidy | interventions — High-Energy Shock Waves

INTERVENTIONS:
Procedure: Ultrasound
Procedure: Serum screen

SUMMARY:
Too much or too little genetic information (chromosome material) can cause abnormal development of the fetus or death. Each year approximately 2.5 million pregnant women are screened for Down Syndrome using invasive screening methods (amniocentesis or chorionic villus sampling). This 11 center study of 38,000 women will compare the accuracy of the several non-invasive tests in the first and second trimesters of pregnancy versus amniocentesis or diagnosis at birth to diagnose aneuploidy or Down Syndrome.

DETAILED DESCRIPTION:
The FASTER (First and Second Trimester Evaluation of Risk) Trial is a multicenter prospective study comparing the accuracy of first and second trimester non-invasive screening methods for Down syndrome and other aneuploidies to diagnosis at delivery or miscarriage/fetal loss). All women will receive the two non-invasive test batteries in both the first and second trimesters. The accuracy of the results of different combinations of non-invasive tests will be compared with diagnosis at delivery or at miscarriage or later fetal loss.

First trimester screening will involve ultrasound measurement of fetal nuchal translucency (NT) thickness at 10-14 weeks gestation, together with maternal age, and serum levels of pregnancy associated plasma protein-A (PPAP-A) and free-beta human chorionic gonadotropin (FbhCG). Second trimester screening will be based on the current standard of care serum "triple screen", which consists of alpha fetoprotein (AFP), unconjugated estriol (uE3), and hCG, performed at 15-18 weeks gestation, together with maternal age and the new serum marker inhibin-A. If patients screen positive (risk >/= 1 in 380), the patients are notified and offered invasive testing at 15 weeks (a serum "quad" test, an additional tube of blood for analysis of the presence of fetal nucleated erythrocytes in maternal blood [NIFTY: National Institute of Child Health and Human Development Fetal Cell Study]), and amniocentesis on those who accept). True positive cases receive counseling. True negative cases, those who decline invasive testing, and those who screen negative after the serum "quad" test, receive routine care with final pediatric outcome. Patients with an a priori risk for Down Syndrome may elect to have invasive fetal testing at 15 weeks after quad testing. For all fetuses with a NT measurement greater than 3 mm, and where karyotype is found to be normal after amniocentesis, will be followed with a repeat ultrasound examination at 18 to 20 weeks gestation, to evaluate fetal anatomy, particularly fetal cardiac structure. Final pediatric examination information will be obtained following delivery. If pregnancy results in miscarriage or later fetal loss, attempts will be made to karyotype any fetal tissue. This is especially important for those pregnancies that abort spontaneously between the time of the first and second trimester methods of screening. Pregnancy outcome data will be obtained in all cases.

ELIGIBILITY:
Inclusion Criteria:

* Women 16 to 45 years old
* Enrolled by participating obstetrical center before 10-14 weeks gestation
* Gestational age 10 weeks three days to 13 weeks six days, with a minimum sonographic crown rump length of 38 mm, maximum 84mm
* Informed consent of patient
* English fluent or accompanied by appropriate interpreter
* Healthy (although co-existing diseases allowed)

Exclusion Criteria:

* Multiple gestation

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38000

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. D'Alton, M. D., Principal Investigator — Columbia-Presbyterian Hospital Medical Center
Locations (10):
- United States (10):
  - University of Colorado Health Sciences Center, Denver, Colorado
  - New England Medical Center, Boston, Massachusetts
  - William Beaumont Hospital Research Institute, Royal Oak, Michigan
  - New York University School of Medicine, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Women and Infants Hospital, Providence, Rhode Island
  - University of Texas Medical Branch, Galveston, Texas
  - University of Utah, Salt Lake City, Utah
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Background] Wald NJ, Kennard A, Hackshaw A, McGuire A. Antenatal screening for Down's syndrome. J Med Screen. 1997;4(4):181-246. doi: 10.1177/096914139700400402. PMID 9494915
- [Background] Wald NJ, Hackshaw AK. Combining ultrasound and biochemistry in first-trimester screening for Down's syndrome. Prenat Diagn. 1997 Sep;17(9):821-9. PMID 9316126
- [Background] Malone FD, D'Alton, MD. Fetal nuchal translucency. Contemporary Obstetrics and Gyncology 1998; 43: 117-31.